CLINICAL TRIAL: NCT06962137
Title: Phase II RAINSPOT: a Multicentric Open Label Trial of Zolbetuximab-Paclitaxel-Ramucirumab in Second Line Setting for CLDN18.2 Positive Gastro-esophageal Adenocarcinoma
Brief Title: Phase II RAINSPOT: Zolbetuximab-Paclitaxel-Ramucirumab for CLDN18.2 Positive Gastro-esophageal Cancer
Acronym: RAINSPOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S70358; ISR007148 (Other Grant/Funding Number: Astellas Pharma Global Development, Inc. (APGD)); 2025-521358-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-24; First posted 2025-05-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic; Gastric Adenocarcinoma and Gastroesophageal Junction Adenocarcinoma
Keywords: Zolbetuximab-Paclitaxel-Ramucirumab; second line; CLDN18.2 positive; gastro-esophageal adenocarcinoma
MeSH Terms: interventions — zolbetuximab

STUDY DESIGN:
Intervention Model Description: The Trial is divided into a prospective open label cohort and a retrospective cohort. There are six participating centers.
  All patients with known CLDN18.2 positivity at baseline are eligible for the prospective cohort, if they did not receive anti-CLD18.2 therapy as first line therapy. It is acceptable to have the CLDN18.2 information tested during their 1st line therapy. All participants who will be included in the trial will remain on the trial until confirmation of disease progression.
  For the retrospective cohort the investigators will identify patients treated with Paclitaxel-Ramucirumab between January 2021 until December 2023 (the era of immunotherapy) in the forementioned centers that have confirmed CLDN18.2 positivity on a baseline biopsy but were not treated with Zolbetuximab in first line setting (nor in experimental setting). Treatment with immunotherapy or targeted therapy in first line setting is allowed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective cohort - Zolbetuximab + SOC Palcitaxel and Ramucirumab (Experimental): * Zolbetuximab: 800 mg/m² loading dose of at C1D1, followed by subsequent doses of 400 mg/m² every 2 weeks. Zolbetuximab should be administered after antiemetic premedication but prior to Paclitaxel-Ramucirumab.
  * Paclitaxel: 80 mg/m² weekly for 3 weeks followed by a week of break according to routine practice.
  * Ramucirumab: 8 mg/kg every 2 weeks according to routine practice.
  Interventions: Drug: zolbetuximab
- Retrospective cohort (Other): For the retrospective cohort the investigators will identify patients treated with Paclitaxel-Ramucirumab between January 2021 until December 2023 (the era of immunotherapy) in the forementioned centers that have confirmed CLDN18.2 positivity on a baseline biopsy but were not treated with Zolbetuximab in first line setting (nor in experimental setting). Treatment with immunotherapy or targeted therapy in first line setting is allowed.
  Interventions: Other: Retrospective cohort, no intervention

INTERVENTIONS:
Drug: zolbetuximab — The investigational product, Zolbetuximab, is a sterile lyophilized powder preparation with the chimeric monoclonal antibody Zolbetuximab as the active pharmaceutical ingredient.
  Arms: Prospective cohort - Zolbetuximab + SOC Palcitaxel and Ramucirumab
Other: Retrospective cohort, no intervention — No intervention
  Arms: Retrospective cohort

SUMMARY:
This study examines whether adding the drug Zolbetuximab to an existing treatment (Paclitaxel and Ramucirumab) can improve patients' survival. The goal is to see if this combination works better for patients whose tumours contain a specific protein (CLDN18.2). The results will be compared to past patient data from those who only received the standard treatment.

Zolbetuximab (Vyloy) is a cancer medicine that is used to treat adults with gastric or gastro-esophageal junction adenocarcinoma (a type of cancer of the stomach or the transition between the stomach and esophagus). Zolbetuximab will be administered via an intravenous infusion in combination with Paclitaxel and Ramucirumab (Cyramza) (two other cancer drugs that are the standard treatment for this condition). Treatment will take place at regular intervals in the hospital. In addition to treatment,patients will undergo a tumour biopsy. While the biopsy procedure may cause some discomfort or pain, it will only be performed if medically justifiable. Patients participation in the study will continue as long as they receive treatment and the disease does not worsen. The overall duration of the study, for all patients, will span several years.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of ICF
2. WHO performance status 0 - 1
3. Histologically proven metastatic gastroesophageal adenocarcinoma
4. Pretreatment with one 1st line therapy according to SOC (+/- immunotherapy)
5. If relapse while adjuvant (immune/chemo) therapy or within 6 months ending adjuvant therapy the adjuvant therapy is considered a first line therapy
6. CLDN18.2-positive (defined as ≥75% of tumour cells showing moderate-to-strong membranous CLDN18.2 staining, as determined by immunohistochemistry using the VENTANA CLDN18 [43-14A] RxDx Assay.
7. Any PDL1 score
8. Use of highly effective methods of birth control
9. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.

Exclusion Criteria:

- 1. Metastatic squamous cell cancer of the esophagus 2. Absolute contra-indication for anti-VEGF inhibitors (tumor perforation, active proteinuria, recent stroke, myocardial infarction, acute arterial thrombosis, active wound problem) 3. Other active malignancy 4. Pretreatment with Zolbetuximab or other anti-CLDN18.2 direct therapy in first line setting once available.

5. Known hypersensitivity to the active substance Zolbetuximab or to any of the excipients [(Arginine, Phosphoric acid (E 338), Sucrose, Polysorbate 80 (E 433)] 6. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive 7. Participation in another interventional Trial with an investigational medicinal product (IMP) or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
OS (overall survival) | From enrollment to the last FU visit of the patient (2 years)
  The primary objective is to evaluate the effect of Zolbetuximab plus Paclitaxel-Ramucirumab on survival in CLDN18.2 positive patients that were previously treated in first line but unexposed to Zolbetuximab or other anti CLDN18.2 targeted therapy.

SECONDARY OUTCOMES:
PFS (progression free survival) | From enrollment till last FU visit of patient (2 years). Data will be reported at the final study report (max 3 years from study start).]
  PFS, which is defined as the time from the date of signature of informed consent until the date of radiological PD (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or death from any cause, whichever is earliest. Patients unprogressed at time of discontinuation for other causes, starting a subsequent line of treatment will be censored for progression at the start of this subsequent treatment.
Safety analysis | Up to 90 days after last Zolbetuximab dose for each individual patient
  Safety analysis. Frequency and severity of treatment emergent AEs, SAEs, irAEs. AEs leading to death,discontinuation of trial intervention

CONTACTS AND LOCATIONS:
Overall Officials: Filip Van Herpe, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (6):
- Belgium (6):
  - UZA, Antwerp
  - Cliniques Universitaires Saint-Luc Brussels, Brussels
  - HUB, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - AZ Delta Roeselare, Roeselare

IPD SHARING:
Plan to Share IPD: No